CLINICAL TRIAL: NCT03782649
Title: Performance Evaluation of a Novel Non-invasive Glucometer, Calibrated Against Validated Interstitial Glucose References
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RSP Systems A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: RSP-08
Record Dates: First submitted 2018-12-03; First posted 2018-12-20 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus
Keywords: Non-invasive glucose monitoring; Raman spectroscopy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RSP-08 (Experimental): All subjects undergo the same procedures. Subjects will be subjected to measurements on the IMD (Working Model 3.4NR), FreeStyle Libre, Dexcom, microdialysis, venous and capillary blood collection.
  Interventions: Device: Working Model 3.4NR

INTERVENTIONS:
Device: Working Model 3.4NR — Investigational Medical Device collecting spectral Raman data from tissue

SUMMARY:
This clinical study has been launched to collect spectral Raman data on the Investigational Medical Device (IMD) compared with reference methods in terms of interstitial fluid samples and capillary and venous references.

DETAILED DESCRIPTION:
Subjects will visit the clinic for a baseline visit and two in-clinic visits. On in-clinic days, subjects will attend the clinic in a fasting state. They will have inserted a Dexcom and Freestyle Libre and a microdialysis catheter. At time = 0, subjects will be administered a glucose rich drink and every 6. minut measurements will be performed. These include a measurement on the IMD, microdialysate, FreeStyle Libre and Dexcom readings. Every 18. minut a venous blood sample will be included and every 36. minut a capillary blood sample will be collected. This continues until time = 180 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18-70 years old
* Patients diagnosed with type 1 or type 2 diabetes (T1D or T2D) (insulin requiring T2D patients)
* Diabetes management strategy: lifestyle regimen + insulin ± oral hypoglycemic agents
* Skin phototype 1-4

Exclusion Criteria:

* For female participants: Pregnancy or subject is attempting to conceive or not willing and able to practice birth control during the study duration
* > 10 cigarettes pr. day
* Participants not able to understand and read Swedish
* In investigator's opinion, participant is not able to follow instructions as specified in the protocol
* Participants not able to hold hand/arm steadily (including tremors and Parkinson's Disease)
* Diagnosed with reduced circulation
* Extensive skin changes, tattoos or diseases on probe application site
* Rejection by screening optical measurements
* Known allergy to medical grade alcohol
* Known allergy to adhesives
* Systemic or topical administration of glucocorticoids for the past 7 days
* Participants undergoing dialysis treatment
* Anti-coagulation or anti-platelet therapy
* Use of beta-blockers
* Medical conditions causing bleeding tendency
* Medical history or any condition that may, in the opinion of the investigator, compromise the subject's ability to participate
* Concomitant medical condition which could present a risk to the safety or welfare of the subject or study staff. Such conditions include but are not limited to HIV and Hepatitis B or C.
* Participants currently enrolled in another study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Generation and validation of prediction models - MARD | One year
  Two in-clinic visits each of a duration of 5-6 hours are scheduled for each subject. Subjects will enter clinic in fasting state and will receive an oral glucose bolus. Glucose excursion is followed with frequent capillary and venous blood samples along with FGM and CGM readings and microdialysis. In parallel, optical glucose data from the investigational medical device will be collected.
  Optical glucose readings will be masked to the subjects.
  Collected data will be used to generate individual calibration models capable of predicting tissue glucose. Models will be validated on independent data sets using Mean Absolute Relative Difference (MARD) endpoint measure.
Generation and validation of prediction models - ISUP | One year
  Two in-clinic visits each of a duration of 5-6 hours are scheduled for each subject. Subjects will enter clinic in fasting state and will receive an oral glucose bolus. Glucose excursion is followed with frequent capillary and venous blood samples along with FGM and CGM readings and microdialysis. In parallel, optical glucose data from the investigational medical device will be collected.
  Optical glucose readings will be masked to the subjects.
  Collected data will be used to generate individual calibration models capable of predicting tissue glucose. Models will be validated on independent data sets using Inter Subject Unified Performance (ISUP) measure.
Generation and validation of prediction models - Consensus Error Grid | One year
  Two in-clinic visits each of a duration of 5-6 hours are scheduled for each subject. Subjects will enter clinic in fasting state and will receive an oral glucose bolus. Glucose excursion is followed with frequent capillary and venous blood samples along with FGM and CGM readings and microdialysis. In parallel, optical glucose data from the investigational medical device will be collected.
  Optical glucose readings will be masked to the subjects.
  Collected data will be used to generate individual calibration models capable of predicting tissue glucose. Models will be validated on independent data sets using Consensus Error Grid Analysis

SECONDARY OUTCOMES:
Evaluation of dynamics between arterial and venous glucose profiles in relation to interstitial glucose levels | One year
  Two in-clinic visits each of a duration of 5-6 hours are scheduled for each subject. Subjects will enter clinic in fasting state and will receive an oral glucose bolus. Glucose excursion is followed with frequent capillary and venous blood samples along with FGM and CGM readings and microdialysis. In parallel, optical glucose data from the investigational medical device will be collected.
  Optical glucose readings will be masked to the subjects.
  A modeling-based evaluation of the dynamics between blood glucose and tissue glucose will be conducted and serve as a secondary endpoint of the study.
Safety evaluation: paucity of adverse events | One year
  Safety will be evaluated in a descriptive manner by the paucity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Per-Anders Jansson, MD, Principal Investigator — Sahlgrenska Universitetssjukhuset, Gothenburg
Locations (1):
- Gothia Forum för Klinisk Forskning, Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No